CLINICAL TRIAL: NCT04050488
Title: Oral Zinc Supplementation Improving Growth and Reducing Morbidity on Very Low Birth Weight Infant
Brief Title: Zinc Supplementation on Very Low Birth Weight Infant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, RismaKK, Principal Investigator, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IKA001
Record Dates: First submitted 2019-07-30; First posted 2019-08-08 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Early-Onset Sepses, Neonatal; Periventricular Haemorrhage Neonatal; Bronchopulmonary Dysplasia; Retinopathy of Prematurity; Enterocolitis, Necrotizing; Small for Gestational Age Infant
MeSH Terms: conditions — Neonatal Sepsis; Bronchopulmonary Dysplasia; Retinopathy of Prematurity; Enterocolitis, Necrotizing | interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled clinical trial in preterm infants (28 - 32 weeks) who are newborn or less than 3 days old who are admitted to the perinatology room. There were two research groups, namely the treatment group (the group that received zinc supplementation) and the control group (the group that received the placebo). In both groups the differences in growth indicators (body weight, body length, and head circumference) will be evaluated, the incidence of morbidity (sepsis, necrotizing enterocolitis, retinopathy of prematurity, intraventricular hemorrhage and bronchopulmonary dysplasia).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization is carried out by research assistants, then making sequential numbers with closed envelopes that have been prepared. The results of the randomization are only known by research assistants. At the age of 3 days or priming> 20cc / kg body weight/day, the research assistant will give a bottle of medicine containing zinc/placebo (according to the results of randomization) without knowing the contents either by the doctor or the room nurse. The researcher monitors all patients who are sampled without knowing which group is the test and which group is the control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Active Comparator): Participants who receive the intervention.
  Interventions: Drug: Zinc Sulfate
- Control Group (Placebo Comparator): Participants who receive the placebo.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Zinc Sulfate — At the age of 3 days or priming> 20cc / kg body weight/day the research assistant will give a bottle of medicine containing zinc (according to the results of randomization) without knowing the contents either by the doctor or the room nurse.
  Arms: Treatment Group
Drug: Placebos — At the age of 3 days or priming> 20cc / kg body weight/day the research assistant will give a bottle of medicine containing placebo (according to the results of randomization) without knowing the contents either by the doctor or the room nurse.
  Arms: Control Group

SUMMARY:
Premature birth is a major cause of neonatal death in addition to neonatal asphyxia and infections.

Early in life, premature babies must get aggressive nutrition so that there is no extrauterine growth restriction (EUGR) in the Intrauterine Growth Restriction (IUGR) group compared to the non-IUGR group.

Other factors that also play a role are long episodes of fasting, the fulfillment of nutrition (macro and micronutrients) from the start, time to start breastfeeding (ASI), duration of parenteral total administration, the incidence of respiratory distress syndrome and incidence of necrotizing enterocolitis.

Zinc is one of the micronutrients which is very risky for deficiency in premature babies.

Babies with zinc deficiency experience growth disorders as much as 67%. In India, infants who received zinc supplementation increased after being given 10 days of zinc supplementation and lower mortality rates in the group with supplementation. Very low birth weight babies and bronchopulmonary dysplasia who received zinc supplementation during the week showed good clinical progress and the growth rate also increased.

The investigators believe this study has the potential for decreasing infant mortality from its current level and can be a growth indicator for preterm babies.

DETAILED DESCRIPTION:
Double-blind randomized controlled clinical trial in preterm infants (28 - 32 weeks) who are newborn or less than 3 days old who are admitted to the perinatology room.

Infant in the intervention group was given elemental zinc supplementation once daily orally compared to placebo in the control group, at 3 days of age until the patient returned home or a maximum of 40 weeks' gestation.

The intervention group was given 10 mg elemental zinc once daily orally compared to placebo in the control group, at 3 days of age and received oral nutrition> 20cc / kg/ day, continued during treatment until the patient returned home or a maximum of 40 weeks' gestation.

Monitored infant development indicators, measured once a week. Monitoring of the incidence of infection in late-onset infants in clinical and laboratory settings according to the existing hospital settings.

The monitoring of NEC events in all research subjects was carried out. Screening ROP at the age of 3 weeks and/or when the baby is going home. The participants were observed to be allowed to go home or a maximum of 40 weeks' gestation if they were still being treated.

ELIGIBILITY:
Inclusion Criteria:

* Preterm (gestational age of 28 - 32 weeks)
* Newborns with a ratio of body weight and gestational age: Small for Gestational Age or Large for Gestational Age
* Get parental approval to be included in the study by signing an informed consent

Exclusion Criteria:

* Newborns with severe congenital abnormalities
* Newborns with digestive tract abnormalities: partial, total obstruction or gastrointestinal atresia
* Newborns with unstable hemodynamic conditions that will affect the survival rate
* Mothers who consume alcohol regularly (≧ 2x a month) during pregnancy
* Newborns with early-onset sepsis

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 364 (Estimated)
Dates: Start 2019-08-20 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Body Weight | 8 to 12 weeks
  Body weight measured by gram
Body Length | 8 to 12 weeks
  Body length measured by centimetres
Head Circumference | 8 to 12 weeks
  Head circumference measured by centimetres

SECONDARY OUTCOMES:
Zinc levels | 8 to 12 weeks
  Determine zinc levels before and after in participants with zinc supplementation and placebo
Rate of mortality | 8 to 12 weeks
  Comparison of mortality rates in participants with zinc supplementation and placebo
Number of participants with side effects | 8 to 12 weeks
  Number of participants with side effects that occur due to zinc supplementation
Number of participants with late-onset sepsis | 8 to 12 weeks
  Comparison of number of participants with late-onset sepsis with zinc supplementation and placebo
Number of participants with intraventricular haemorrhage | 8 to 12 weeks
  Comparison of number of participants with intraventricular haemorrhage with zinc supplementation and placebo
Number of participants with bronchopulmonary dysplasia | 8 to 12 weeks
  Comparison of number of participantswith bronchopulmonary dysplasia with zinc supplementation and placebo
Number of participants with retinopathy of prematurity | 8 to 12 weeks
  Comparison of number of participantswith retinopathy of prematurity with zinc supplementation and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Henri Azis, Master, Principal Investigator — Fakultas Kedokteran Universitas Indonesia

IPD SHARING:
Plan to Share IPD: No
This research can be done in other places by considering the condition of existing medical servants. When giving a good outcome, you can contact the research contact

REFERENCES:
- [Background] Terrin G, Berni Canani R, Passariello A, Messina F, Conti MG, Caoci S, Smaldore A, Bertino E, De Curtis M. Zinc supplementation reduces morbidity and mortality in very-low-birth-weight preterm neonates: a hospital-based randomized, placebo-controlled trial in an industrialized country. Am J Clin Nutr. 2013 Dec;98(6):1468-74. doi: 10.3945/ajcn.112.054478. Epub 2013 Sep 11. PMID 24025633
- [Background] Banupriya N, Bhat BV, Benet BD, Catherine C, Sridhar MG, Parija SC. Short Term Oral Zinc Supplementation among Babies with Neonatal Sepsis for Reducing Mortality and Improving Outcome - A Double-Blind Randomized Controlled Trial. Indian J Pediatr. 2018 Jan;85(1):5-9. doi: 10.1007/s12098-017-2444-8. Epub 2017 Sep 11. PMID 28891027